CLINICAL TRIAL: NCT01302340
Title: Two Phase, Repeated Crossover Study With Dose Escalation on Delta(9)-Tetrahydrocannabinol (Delta-THC) in Behavioral Disturbances in Dementia
Brief Title: Delta-THC in Behavioral Disturbances in Dementia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: European Union (Other)
Responsible Party: Principal Investigator, Marcel Olde Rikkert, Prof. dr., Radboud University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GER001-02-01; 2009-019329 (Other Grant/Funding Number: Province of Gelderland&Overijssel); 2010-024577-39 (EudraCT Number); Supplies Investigational Drug (Other Grant/Funding Number: Echo pharmaceuticals)
Record Dates: First submitted 2011-02-10; First posted 2011-02-24 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Dementia
Keywords: Dementia; Alzheimer; Cannabis; THC; Behavioral Disturbances; Neuropsychiatric Inventory
MeSH Terms: conditions — Dementia; Marijuana Abuse; Mental Disorders | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Delta-THC (Active Comparator): THC will be administered twice daily during three consecutive days per treatment block(0.75 or 1.5 mg twice daily)
  Interventions: Drug: Delta-THC
- placebo (Placebo Comparator): Placebo will be administered twice daily during three consecutive days per treatment block.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Delta-THC — Active treatment consists of THC in tablet form. Patients receive 0.75 mg THC twice daily during the first three treatment blocks (period A) and 1.5 mg THC twice daily during the latter three treatment blocks (period B). Placebo treatment consists of two tablets daily and is matched to the active treatment for taste, color and size. Study medication will be administered at 10 a.m. and 4 p.m., by the primary caregiver. These time points are chosen because NPS often occur later on the day, when fatigue and external signals build up to the stress and result in NPS. The order of administration of THC and placebo (1:1) will be determined by randomization per block: THC followed by placebo or placebo followed by THC.
  Other Names: Namisol; Cannabis; ECP002A
  Arms: Delta-THC
Drug: placebo — Active treatment consists of THC in tablet form. Patients receive 0.75 mg THC twice daily during the first three treatment blocks (period A) and 1.5 mg THC twice daily during the latter three treatment blocks (period B). Placebo treatment consists of two tablets daily and is matched to the active treatment for taste, color and size. Study medication will be administered at 10 a.m. and 4 p.m., by the primary caregiver. These time points are chosen because NPS often occur later on the day, when fatigue and external signals build up to the stress and result in NPS. The order of administration of THC and placebo (1:1) will be determined by randomization per block: THC followed by placebo or placebo followed by THC.
  Other Names: Placebo Namisol
  Arms: placebo
Drug: Delta-THC — In case either 2 times daily 1 tablet 0,75mg or 2 times daily 1 tablet 1.5mg Delta-THC appeared to be efficacious for a particular patient, this patient can continue the effective dose of delta-THC in an open label extension phase during 6 months.
  Other Names: Namisol; Cannabis; ECP002A
  Arms: Delta-THC

SUMMARY:
Dementia is a common chronic condition, with predicted increasing prevalence. Nearly all patients with dementia will experience neuropsychiatric symptoms (NPS). This causes significant burden for the individual patients and their caregivers. Current treatment has only modest efficacy and important side-effects. Formulations with Δ9-tetrahydrocannabinol (THC), the psycho-active compound of cannabis, are currently being registered for spasms in multiple sclerosis and other diseases, and may have beneficial effects on NPS.

DETAILED DESCRIPTION:
Design Phase II pilot study, multi-center, repeated cross-over, double blinded randomized trial. The study consists of two weeks baseline measurements to assure that the neuropsychiatric symptoms are stable and six successive treatment blocks of 2 weeks. Each treatment block lasts for two weeks and contains two double-blinded drug periods, each lasting three days of oral THC or placebo, separated by four day washout periods. After three treatment blocks (period A), the dosage of active treatment was increased for the latter three treatment blocks (period B). After the two treatment periods, subjects will proceed to the extension phase if applicable.

Study centers The department of Geriatrics from Radboud University Nijmegen Medical Centre and the department of Elderly from Vincent van Gogh voor Geestelijke Gezondheidszorg Venray (VVG) will participate in this multi center study.

Participants 20 subjects with dementia and NPS. Intervention Namisol® in doses of twice daily 0,75 mg tablet (period A) and twice daily 1.5 mg (period B) THC oral tablets. Placebo of twice daily 0,75 mg and twice daily 1.5 mg oral tablets Outcome measures Primary outcome is NPI score, secondary CMAI, Zarit Burden scale. Other outcomes include vital signs, side-effects, physical exam, mobility and pharmacogenetics.

Visits This study will be assessed fully ambulatory, starting with a 5 hour clinical visit on day 1 and 8 of block 1 and a phone call on day 2 and 9 for assessment of Adverse Events. Furthermore, the research physician will conduct a weekly home visit weekly during the crossover phase for assessment of , among others, the primary outcome measure. These visits will all be repeated in period B of the crossover phase.

During the 6 month open label extension phase, subjects will visit the clinic three times.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Alzheimer's Disease (AD), Vascular Dementia (VD) or mixed, according to the criteria of NINCDS-ADRDA or NINCDS-AIREN
* Clinical Dementia Rating score between 0.5 and 3
* NPS symptoms, with at least agitation or aggression

Exclusion Criteria:

* Diagnosis of Lewy Body Dementia (LBD) or Fronto-Temporal Dementia (FTD)
* Major psychiatric disorder
* Severe concomitant illness, seizure, arrhythmias (except sinus arrhythmia and atrial fibrillation), heart failure New York Heart Association (NYHA) class III or IV
* Tri Cyclic Antidepressives (TCA) or opioids used within 30 days before randomization till the end of the study
* Changes in dosage of antidepressives within 6 weeks before randomization and during study, and changes in dosage antipsychotics or benzodiazepines within 2 weeks prior to randomization and during study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Neuropsychiatric Inventory (NPI) | At day 3 and 10 during treatment blocks and after 1 month, 3 months and 6 months in the open label extension phase
  Improvement in behavior compared to placebo is measured with the NPI, which is the standard measure of Neuro Psychiatric Symptoms in most clinical trials.

SECONDARY OUTCOMES:
Cohen-Mansfield Agitation Inventory (CMAI) | At days 1, 3, 8, and 10 during treatment blocks 1 and 4 and weekly during treatment blocks 2, 3, 5 and 6 and months 1, 3, 6 and 6 during extension phase
  Improvement in agitation compared to placebo and during long term treatment is measured with CMAI. It is useful in determining fluctuations in behaviors and emotional states in Alzheimer's Disease
Zarit Burden Scale (ZBS) | At days 3 and 10 during treatment blocks and months 1, 3 and 6 during extension phase
  Reducing caregiver stress compared to placebo and during long term treatment by focusing on the patients' behavior compared to Zarit burden interviews with the caregiver.
Visual Analogue Scale (VAS) Bowdle for feeling high | At days 1, 3, 8, and 10 during treatment blocks 1 and 4 and weekly during treatment blocks 2, 3, 5 and 6 and months 1, 3, 6 and 6 during extension phase
  severity and duration of feeling high episodes
Gait rite® | At days 1 and 8 during blocks 1 and 4 and at 1, 3 and 6 months during extension phase
  Improvement and/or safety compared to placebo and during long term treatment on balance and mobility. It is a non invasive and highly feasible mobility assessment.
Sway Star® | At days 1 and 8 during blocks 1 and 4 and at 1, 3 and 6 months during extension phase
  Improvement and/or safety compared to placebo and during long term treatment on balance and mobility. It is a non invasive and highly feasible mobility assessments.
Time up and go | At days 1, 3, 8, and 10 during treatment blocks 1 and 4 and weekly during treatment blocks 2, 3, 5 and 6 and months 1, 3, 6 and 6 during extension phase
  Improvement and/or safety compared to placebo and during long term treatment on balance and mobility in elderly patients.
Tinetti Balance Assessment Tool | At days 1, 3, 8, and 10 during treatment blocks 1 and 4 and weekly during treatment blocks 2, 3, 5 and 6 and months 1, 3, 6 and 6 during extension phase
  Improvement and/or safety compared to placebo and during long term treatment on balance and mobility in elderly patients. It is a performance-oriented assessment of mobility problems in elderly patients.
pharmacogenetics | day 1
  The following polymorphisms will be genotyped:
  * CYP2C9*2
  * CYP2C9*3
  * CYP2C19*2
  * CYP2C19*3
  * CYP2C19*17
  To investigate the role of CYP2C9 and CYP2C19 genetic polymorphisms in the interindividual variation in pharmacokinetics, efficacy and adverse events of THC.

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Olde Rikkert, prof MD, Principal Investigator — Radboud University Medical Center
Locations (2):
- Netherlands (2):
  - Radboud university medical center, Nijmegen, Gelderland
  - Vincent van Gogh Institute for Psychiatry, department of Elderly, Venray, Limburg

REFERENCES:
- [Derived] Bosnjak Kuharic D, Markovic D, Brkovic T, Jeric Kegalj M, Rubic Z, Vuica Vukasovic A, Jeroncic A, Puljak L. Cannabinoids for the treatment of dementia. Cochrane Database Syst Rev. 2021 Sep 17;9(9):CD012820. doi: 10.1002/14651858.CD012820.pub2. PMID 34532852